CLINICAL TRIAL: NCT01280539
Title: The Effect of Transcutaneous Electrical Nerve Stimulation (TENS) in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Provinciale Hogeschool Limburg (Other)
Responsible Party: Principal Investigator, Koen Cuypers, Drs, Hasselt University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MECU2012-002
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Transcutaneous electrical nerve stimulation; Cortical Excitability
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TENS (Experimental): Transcutaneous electrical nerve stimulation will be applied on the impaired hand
  Interventions: Device: Transcutaneous electrical nerve stimulation
- Sham TENS (Sham Comparator): Sham TENS will be applied to the impaired hand
  Interventions: Device: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — 3 weeks, 5 times a week, 60 minutes a day.

SUMMARY:
In this study the researchers want to investigate the effects of long-term transcutaneous electrical nerve stimulation on the cortical excitability of persons with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Expanded Disability Status Scale (EDSS) scores between 2 and 6.5
* Stable MS (no relapse during the last 3 months before study onset)
* sensory impairment
* age: between 18 and 68 years old

Exclusion Criteria:

- Patients with other pathologies associated with peripheral and/or central sensory dysfunction or under psychotropic or antiepileptic medication

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in cortical excitability | Baseline, immediately after and 3 weeks after the intervention
  Cortical excitability will be assessed using transcranial magnetic stimulation (TMS)

CONTACTS AND LOCATIONS:
Locations (1):
- Hasselt University (BIOMED), Diepenbeek, Limburg, Belgium